CLINICAL TRIAL: NCT02244957
Title: Right Ventricular Hemodynamics Using Cardiac Magnetic Resonance Imaging in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Obstructive Sleep Apnea (OSA)
Brief Title: Right Ventricular Hemodynamics Using Cardiac MRI in Patients COPD and OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Robert L. Owens, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD140959
Record Dates: First submitted 2014-09-15; First posted 2014-09-19 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea; Chronic Obstructive Pulmonary Disease; Overlap Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bi-level positive airway pressure (BPAP) (Active Comparator): Bi-level positive airway pressure (BPAP)
  Interventions: Device: Bi-level positive airway pressure (BPAP)
- Nocturnal oxygen (Active Comparator): Nocturnal oxygen
  Interventions: Drug: Nocturnal oxygen

INTERVENTIONS:
Device: Bi-level positive airway pressure (BPAP) — Overlap patients randomized to BPAP will be titrated as per American Academy of Sleep Medicine (AASM) guidelines and oxygen if needed based on saturations <88% while on stable bi-level settings.
  Other Names: BPAP
  Arms: Bi-level positive airway pressure (BPAP)
Drug: Nocturnal oxygen — Oxygen will be titrated to keep resting oxygen saturation (as measured by pulse oximeter) more than 88 percent. The duration of therapy will be six months.
  Other Names: NOT
  Arms: Nocturnal oxygen

SUMMARY:
The coexistence of chronic obstructive pulmonary disease (COPD) and obstructive sleep apnea (OSA) in the same patient has been termed overlap syndrome, affecting 1% of the U.S. population.The investigators propose to conduct this study that aims: (1) to compare right and left ventricular hemodynamic parameters using cardiac magnetic resonance imaging (MRI) in overlap syndrome vs. COPD only and OSA only; (2) to compare the effects of bi-level positive airway pressure (BPAP) vs. nocturnal oxygen therapy (NOT) on right ventricular (RV) hemodynamics in overlap syndrome.

This study will allow us to test the hypothesis: (1) Patients with overlap syndrome have more RV dysfunction than those with COPD only or OSA only; (2) treatment of both hypoxemia and hypercapnia during sleep will improve RV hemodynamics compared with treatment of hypoxemia alone in patients with overlap syndrome.

DETAILED DESCRIPTION:
Despite the high prevalence of overlap syndrome, few data are available on its pathophysiology and clinical consequences of these patients. Overlap syndrome has recently been reported to have excess cardiovascular mortality compared with COPD alone. However, no study has evaluated the mechanisms of excess cardiovascular mortality in untreated overlap syndrome. In addition, no prospective, randomized, controlled data are currently available on treatment of overlap syndrome.

This study is divided into two parts. The first part (Part 1) is a cross-sectional cohort study comparing subjects with overlap syndrome to those with COPD alone and those with OSA alone. Patients with COPD and OSA overlap syndrome will be evaluated by an overnight sleep study, cardiac MRI, serum inflammatory biomarker, urine catecholamine level, pulmonary function test, and questionnaires of sleep and health related quality of life. These measurement will be compared between overlap syndrome and control groups with either COPD or OSA alone.

The second part (Part 2) of the study is a prospective, parallel-group, randomized, controlled pilot study examining the effect of BPAP (and nocturnal oxygen if needed) vs. nocturnal oxygen therapy alone in patients with overlap syndrome (20 subjects in each treatment arm). The same measurement done during Part 1 will be repeated to evaluate the treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women with age more than 18 years.
* Known diagnosis of stable COPD (GOLD stage 2 or higher) or OSA.

Exclusion Criteria:

* Already using continuous positive airway pressure (CPAP), BPAP device, or nocturnal oxygen.
* Known or suspected renal failure with estimated Glomerular filtration (GFR) <50 ml/min/1.73 m2 or serum creatinine > 1.5 mg/dl.
* Chronic atrial fibrillation or frequent premature ventricular contraction (> 10 beats per hour)
* Women known to be pregnant or planning to be pregnant in next 6 months.
* Known contraindication to MRI: cardiac pacemaker, metallic heart valves, metallic implants, history of claustrophobia.
* If taking sildenafil or related drugs, unable to stop it within 48 hours of the study visit.
* Uncontrolled COPD or acute COPD exacerbation.
* Unstable cardiac diseases.
* Known chronic inflammatory diseases like lupus or active infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Owens, MD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Obstructive Pulmonary Disease (COPD): Subjects with only Chronic Obstructive Pulmonary Disease (COPD)
- Overlap Syndrome: Subjects with simultaneous Obstructive Sleep Apnea (OSA) and Chronic Obstructive Pulmonary Disease (COPD). The dual diagnosis of these two conditions is referred to as Overlap Syndrome.
Period: Overall Study
Arm/Group | Chronic Obstructive Pulmonary Disease (COPD) | Overlap Syndrome
Started | 7 | 16
Completed | 6 | 16
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: one subject was dropped due to lack of efficacy
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Obstructive Pulmonary Disease (COPD) | Overlap Syndrome | Total
Number analyzed (Participants) | 6 | 16 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.4) | 63.5 (4.2) | 63.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 14 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 5 | 13 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 16 | 22

OUTCOME MEASURES:

1. Primary Outcome: Right Ventricular Remodeling Index
Description: Defined as the ratio between RVMI and RV end-diastolic volume index using MRI
Time Frame: Six months
Population: one subject was dropped due to lack of efficacy
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Chronic Obstructive Pulmonary Disease (COPD) | Overlap Syndrome
Number analyzed (Participants) | 6 | 16
ratio | 0.3747 (0.06335) | 0.2817 (0.03630)

2. Secondary Outcome: Right Ventricular Mass Index
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Right Ventricular End Systolic and Diastolic Volume
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Right Ventricular Ejection Fraction
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Myocardial Extracellular Volume
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Left Ventricular Remodeling Index
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Left Ventricular Mass Index
Description: MRI
Time Frame: Six months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Left Ventricular End Systolic and Diastolic Volume
Description: MRI
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Left Ventricular Ejection Fraction
Description: MRI
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Serum C-reactive Protein Level
Description: blood test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Serum Tumor Necrosis Factor-alpha Level
Description: blood test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Serum Interleukin-6 Level
Description: blood test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Serum Intercellular Adhesion Molecule-1
Description: blood test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Serum P-selectin Level
Description: Blood test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Urine Catecholamine Level
Description: Urine test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: 6 Minute Walk Distance
Description: Low-grade physical activity test
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Quality of Life Score Through St. George's Respiratory Questionnaire (SGRQ)
Description: Questionnaire
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Degree of Daytime Sleepiness Through Epworth Sleepiness Scale (ESS)
Description: Questionnaire
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Sleep Quality Through Pittsburgh Sleep Quality Index (PSQI)
Description: Questionnaire
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: General Health Status Through Short Form 36 (SF-36) Health Survey
Description: Questionnaire
Time Frame: 6 months
Population: No data collected as study was terminated prior to randomization
Arm/Group | Bi-level Positive Airway Pressure (BPAP) | Nocturnal Oxygen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Chronic Obstructive Pulmonary Disease (COPD) | Overlap Syndrome
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/16
Other Adverse Events (participants affected / at risk) | 0/7 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT02244957/Prot_000.pdf